CLINICAL TRIAL: NCT01838330
Title: Effects of High Dietary Fiber Supplementation on Uremic Retention Molecules and Inflammation in Diabetic Chronic Kidney Disease (CKD)
Brief Title: Effects of High Dietary Fiber Supplementation in Diabetic Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Srinvasan Beddhu, MD, Faculty Sponsor, University of Utah
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB_00052609
Record Dates: First submitted 2013-01-30; First posted 2013-04-24 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Kidney Disease
Keywords: Kidney Disease; Fiber; Dietary Intervention
MeSH Terms: conditions — Kidney Diseases | interventions — Psyllium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chronic Kidney Disease Stage 3-4 (Experimental): Study participants with stage 3 or 4 CKD will receive 15 grams/day of soluble fiber psyllium for the first week, followed by 30 grams/day of a soluble fiber psyllium for 4 months.
  Interventions: Dietary Supplement: psyllium
- Chronic Kidney Disease Stage 1-2 (No Intervention): Study participants with stage 1 or 2 CKD will not receive study treatment

INTERVENTIONS:
Dietary Supplement: psyllium — 15 grams/day for 1 week, followed by 30 grams/day for 4 months
  Other Names: Metamucil
  Arms: Chronic Kidney Disease Stage 3-4

SUMMARY:
Loss of kidney function results in accumulation in the blood of molecules that are either excreted or metabolized by the kidney. Collectively, these molecules are termed Uremic Retention Molecules (URMs) or toxins. It is increasingly recognized that colonic bacterial metabolites like p-cresyl sulfate and indoxyl sulfate that are absorbed from the colon and excreted by the kidney may contribute to the pool of compounds implied in uremic toxicity. Indeed, these URMs have been linked to increased levels of inflammation markers, chronic kidney disease (CKD) progression, cardiovascular disease and overall mortality in CKD and/ or hemodialysis patients. Therefore, interventions that target the production or absorption of URMs from the gut might decrease inflammation and oxidative stress that are commonly seen in the uremic milieu. The National Health and Nutrition Examination Survey III (NHANES III) data show that high dietary fiber intake is associated with decreased serum levels of C-reactive protein (CRP) in those with and without CKD and these associations are much stronger in the CKD population. A possible explanation of this effect is that a high fiber diet in CKD patients modulates the bacterial production, intestinal absorption and finally the serum levels of URMs like p-cresyl sulfate and indoxyl sulfate, which in turn results in decrease in inflammation.

OBJECTIVES:

Hypothesis:

1. Higher serum levels of markers of inflammation such as high sensitivity C-reactive protein (hsCRP), interleukin 6 (IL-6) and tumor necrosis factor (TNF) -α seen in stage 4 CKD (estimated Glomerular Filtration Rate 15-29 ml/min/1.73 m2) compared to stage 2 CKD (estimated Glomerular Filtration Rate 60-89 ml/min/1.73 m2) is partly explained by the higher circulating levels of URMs (p-cresyl sulfate and indoxyl sulfate) in stage 4 CKD, and
2. Dietary supplementation in stage 4 CKD with 30g/d of a soluble fiber Psyllium (brand name-Metamucil TM) will decrease circulating URMs levels and thereby, decrease serum levels of inflammation markers and urinary levels of transforming growth factor (TGF)-β, a marker of kidney fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with or without diabetes and Stage 1 or 2 CKD (estimated Glomerular Filtration Rate > 60 mL/min/1.73 m2) with urine dipstick positive for protein or urinary albumin/ creatinine > 30 mg/g of creatinine; or
* Stage 3 or 4 CKD (estimated Glomerular Filtration Rate < 60 to 15 mL/min/1.73 m2).

Exclusion Criteria:

* Pregnant women
* Prisoners
* Bowel obstruction
* Enrolled in other interventional studies.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
p-cresyl sulfate serum concentration | 4 months
  Comparison of serum p-cresyl sulfate concentration between Stage 3-4 CKD subjects (following treatment with soluble fiber psyllium) and Stage 1-2 CKD subjects (having received no study treatment)

SECONDARY OUTCOMES:
Indoxyl sulfate serum concentration | 4 months
  Comparison of serum indoxyl sulfate concentration between Stage 3-4 CKD subjects (following treatment with soluble fiber psyllium) and Stage 1-2 CKD subjects (having received no study treatment)
Interleukin-6 (IL-6) serum concentration | 4 months
  Comparison of serum IL-6 concentration between Stage 3-4 CKD subjects (following treatment with soluble fiber psyllium) and Stage 1-2 CKD subjects (having received no study treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Nestor Almeida, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah nephrology clinics, the internal medicine and endocrinology clinics, Salt Lake City, Utah, United States